CLINICAL TRIAL: NCT00269659
Title: Serial Evaluation of Left Bundle Branch Block; Role of New Imaging Techniques. Three-Dimensional Echocardiography, Tissue Doppler Imaging, and Magnetic Resonance Imaging
Brief Title: Evaluating Effects of a Left Bundle Branch Block
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: The Interuniversity Cardiology Institute of the Netherlands (Other Government)
Other Study IDs: VUMC 2003/147
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Mechanical Dyssynchrony; Heart Failure; Bundle-Branch Block
Keywords: Left Bundle Branch Block; Regional cardiac function; Global cardiac function; Mechanical asynchrony; Echocardiography; 2D echocardiography; Tissue Doppler Imaging; Real-time 3D echocardiography; Cardiovascular Magnetic Resonance Imaging-tagging
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A left bundle branch block (LBBB) is related to abnormal cardiac conduction and mechanical asynchrony and is associated with hypertension and coronary artery disease. Improved evaluation of left ventricular (LV) mechanical asynchrony is needed, because of the increasing number of patients with a LBBB and heart failure. A variety of patterns of mechanical activation can be observed in LBBB patients.

Novel imaging modalities such as tissue Doppler imaging, real-time 3D echocardiography and cardiovascular magnetic resonance imaging provide information about regional and global LV function in healthy subjects, patients without a LBBB with heart failure, patients with a LBBB without heart failure, and patients with a LBBB with heart failure.

The investigators want to evaluate the different patient groups with the novel imaging modalities and they want to compare the novel imaging modalities with each other.

The investigators hypothesized that, between the groups, differences concerning regional and global LV function are measurable.

Each novel imaging technique has its own advantages and limitations but are comparable in measuring regional and global LV function.

DETAILED DESCRIPTION:
Within a time period of 3 years we evaluate different groups of patients and measure regional and global cardiac function.

Therefore, we developed an echocardiography screening-protocol in which we use conventional 2D echocardiography and conventional Doppler echocardiography, extended with tissue Doppler imaging and real-time 3D echo acquisitions.

In a limited group of patients we perform a specially designed cardiovascular magnetic resonance imaging protocol which uses artificially induced grid-lines to evaluate regional and global cardiac function.

Patients are referred to our hospital because of evaluation of their LBBB and or heart failure. We ask them if they would like to undergo the echocardiography and the cardiovascular magnetic resonance imaging.

After a year we want to repeat the measurements in a small group of the patients to re-evaluate regional and global cardiac function.

All patients should have a sinus rhythm and adequate acoustic windows. Patients should not have contraindications for cardiovascular magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-85 years
* Left bundle branch block with or without heart failure
* Narrow QRS duration with or without heart failure

Exclusion Criteria:

* No informed consent
* No sinus rhythm
* Poor acoustic window
* For cardiovascular magnetic resonance imaging part:

  * claustrophobia
  * devices

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2004-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Otto Kamp, MD, PhD, Study Chair — Amsterdam UMC, location VUmc
Locations (1):
- VU Medical Center, Amsterdam, Netherlands